CLINICAL TRIAL: NCT06277648
Title: Comparison of the Pericapsular Nerve Group (PENG) and Suprainguinal Fascia Iliaca Blocks (SIFIB) in Elderly Patients With Subtrochanteric Femur Fractures
Brief Title: the Pericapsular Nerve Group (PENG) and Suprainguinal Fascia Iliaca Blocks (SIFIB) in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 18-2021
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Collum Femoris Fracture; Pericapsular Nerve Group Block; Suprainguinal Fascia Iliaca Block
Keywords: femur fracture; suprainguinal fascia iliaca block; pericapsular nerve group block; elderly patients; postoperative pain
MeSH Terms: conditions — Femoral Fractures; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: a double-blind, prospective, randomized, controlled study
Who Masked: Participant, Outcomes Assessor
Masking Description: The orthopaedic surgeon responsible for the study was blinded to the study groups. This surgeon was the sole evaluator of postoperative pain scores and total analgesia consumption.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): All patients received standard spinal anaesthesia procedures with multimodal pain protocol postoperatively.
- PENG block (Experimental): All patients received standard spinal anaesthesia procedures with PENG block postoperatively.
  Interventions: Procedure: PENG block
- SIFI block (Experimental): All patients received standard spinal anaesthesia procedures with SIFIB postoperatively.
  Interventions: Procedure: SIFIB

INTERVENTIONS:
Procedure: PENG block — PENG block was performed by the primary investigator (B.C) following proper skin disinfection with the patient in the supine position. Under the guidance of a low-frequency curvilinear ultrasound probe, the iliopubic eminence and the psoas tendon were identified, and local anaesthetic as 30 mL 0.375% bupivacaine was injected between the periosteum and psoas tendon following negative aspiration.
  Other Names: pericapsuşar nerve group block
  Arms: PENG block
Procedure: SIFIB — The high-frequency linear probe was placed medial to the anterosuperior iliac spine in a parasagittal orientation to visualize the bow tie appearance formed by the sartorius's internal oblique and iliacus muscles. The needle tip was placed under fascia iliaca through an in-plane approach, and local anaesthetic as 30 mL 0.375% bupivacaine was injected from the caudad to the cephalic direction.
  Other Names: suprainguinal fascia iliaca block
  Arms: SIFI block

SUMMARY:
This clinical trial aims to compare the effect of the pericapsular nerve group (PENG) and suprainguinal fascia iliaca blocks (SIFIB) on pain management in elderly patients with subtrochanteric femur fractures.

The participants will be patients determined to have proximal femoral nailing. According to randomisation, each participant will receive either PENG or SIFIB postoperatively after spinal anaesthesia. The investigator will measure postoperative pain scores, total amount of analgesic consumption and motor ability postoperatively.

DETAILED DESCRIPTION:
Randomization and blindness Randomization was designed as 3 (n= 25) named Groups A, B, and C in a 1:1:1 ratio with a computer-based algorithm and sealed in opaque envelopes by the surgeon assigned to the study. The investigator anesthesiologist selected an envelope in order of numbers written on it and proceeded with PENG if it was Group A and SIFIB if it was Group B. There was no other intervention than intravenous analgesia if it was Group C. The orthopaedic surgeon responsible for the study was blinded to the study groups. This surgeon was the sole evaluator of postoperative pain scores and total analgesia consumption. All block procedures were performed by the primary investigator (B.C.) The duration of block performance and number of needle manipulations before local anaesthetic injections were recorded by the anaesthesia technician assisting the procedure.

Anaesthesia, interventions, and post-interventional follow-up Standardization All patients received standard spinal anaesthesia procedures with 10 mg of heavy Marcaine (2 mL of bupivacaine 0.5%) and 20 µg of fentanyl (0.5 ml) at L3-4 intervertebral space with the aid of midazolam 0.02 mg /kg and ketamine 0.3 mg/kg to-analgesia to achieve sitting position. According to randomization, patients in the study groups (Group PENG and SIFIB) received block procedures with the same local anaesthetic mixture as 30 mL 0.375% bupivacaine postoperatively in the recovery room under monitorization. The same analgesia plan was ordered for all participants as paracetamol 1 gr (four times daily), tenoxicam 20 mg (daily) and dexamethasone 8 mg once postoperatively. They received rescue analgesia only if they had persistent pain scores higher than 4 of 10 or asked for analgesia, as 1mg/kg tramadol (maximum daily dose, 4x1).

Interventions; block procedures PENG block was performed by the primary investigator (B.C) following proper skin disinfection with the patient in the supine position. Under the guidance of a low-frequency curvilinear ultrasound probe, the iliopubic eminence and the psoas tendon were identified, and local anaesthetic was injected between the periosteum and psoas tendon following negative aspiration.

For SIFIB, the high-frequency linear probe was placed medial to the anterosuperior iliac spine in a parasagittal orientation to visualize the bow tie appearance formed by the sartorius internal oblique and iliacus muscle. The needle tip was placed under fascia iliaca through an in-plane approach, and local anaesthetic was injected from the caudad to the cephalic direction.

Outcome Measures Primary outcome The primary outcome of this study is the pain scores. They were assessed by the same orthopaedic surgeon using the NRS (which ranges from 0 to 10, where zero represents the absence of pain, and 10 signifies the worst imaginable pain) at postoperative intervals of 0,4, 8, 12, and 24 hours.

Secondary outcomes The blinded orthopaedic surgeon recorded the number of times rescue analgesia was applied within 24 hours postoperatively as analgesic consumption. Also, block performances were compared by the duration of interventions and the presence of motor block as hip adduction at the postoperative 6th hour.

Sample size and statistical analysis The sample size was based on detecting a change of 2 units or more in mean pain scores (the primary outcome) using analysis of covariance on the outcomes at the follow-up time point. Using an estimated standard deviation of 2 units for pain scores (0-10) with standard type I and type II error rates, we calculated that 20 patients per group would be needed. To allow dropouts or exclusions, we enrolled 25 patients on each group to have a total sample size of 75 participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65
* Patients scheduled for proximal femoral nailing
* Patients with American Society of Anesthesiologists (ASA) Physical Status classification of I to IV.

Exclusion Criteria:

* refusal to participate
* a history of neurological deficits or neuropathy
* infection at the site of block application
* coagulopathy
* allergy to local anaesthetics
* patients with severe cardiopulmonary insufficiency or renal impairment
* mental illness.
* prolonged surgery due to orthopaedic complications of more than 3 hours, necessitating conversion of spinal anaesthesia to general anaesthesia.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
pain scores | postoperative 24 hour
  the numeric rating scale (which ranges from 0 to 10, where zero represents the absence of pain, and 10 signifies the worst imaginable pain)

SECONDARY OUTCOMES:
rescue analgesia | postoperative 24 hour
  The number of times rescue analgesia was applied

CONTACTS AND LOCATIONS:
Overall Officials: Berna Caliskan, Principal Investigator — Haseki Training and Research Hospital Anesthesiology and Reanimation Department
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Sultangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vamshi C, Sinha C, Kumar A, Kumar A, Kumari P, Kumar A, Kumar S, Arun SK. Comparison of the efficacy of pericapsular nerve group block (PENG) block versus suprainguinal fascia iliaca block (SFIB) in total hip arthroplasty: A randomized control trial. Indian J Anaesth. 2023 Apr;67(4):364-369. doi: 10.4103/ija.ija_311_22. Epub 2023 Apr 10. PMID 37303868
- [Background] Aliste J, Layera S, Bravo D, Jara A, Munoz G, Barrientos C, Wulf R, Branez J, Finlayson RJ, Tran Q. Randomized comparison between pericapsular nerve group (PENG) block and suprainguinal fascia iliaca block for total hip arthroplasty. Reg Anesth Pain Med. 2021 Oct;46(10):874-878. doi: 10.1136/rapm-2021-102997. Epub 2021 Jul 20. PMID 34290085